CLINICAL TRIAL: NCT03311815
Title: A COMPREHENSIVE AND RAPID DIAGNOSIS PLATFORM OF PERSONALIZED MEDICINE FOR THE TREATMENT OF ACUTE MYELOID LEUKEMIA. PROSPECTIVE, MULTICENTER AND NON-INTERVENTIONAL STUDY
Brief Title: Diagnostic Platform to Perform Centralized and Standardized Rapid Molecular Diagnosis by Next Generation Sequencing (NGS) in Patients Diagnosed With Acute Myeloid Leukemia.
Status: Completed | Type: Observational
Sponsor: PETHEMA Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: NGS-LMA
Record Dates: First submitted 2017-10-04; First posted 2017-10-17 (Actual); Last update posted 2021-02-16 (Actual); Status verified 2021-02

CONDITIONS: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — bone marrow and peripheral blood samples from AML patients
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: NGS techniques — Using NGS techniques we will detect the recurrently mutated genes in AML to establish the biological role of each mutation

SUMMARY:
NGS studies will be done in stem cell leukemic population. The analysis of the samples to the diagnosis will be carried out using the 26 consensus genes: ASXL1 had, CBL, CEBPA, DNMT3A, EZH2, FLT3, GATA2, IDH1, IDH2, JAK2, KIT, KRAS, MPL, MLL, NPM1, NRAS, PTPN11, RUNX1, SETBP1, SF3B1, SRSF2, TET2, TP53, U2AF1, WT1. Regarding the 26 genes panel, it would have the advantage that the quantification of DNA from each sample will be carried out by fluorimetry using the AmpliSeq or TruSeq on Ion platforms torrent Proton or MySeq are handled in different laboratories.

Using NGS techniques the investigator will detect the recurrently mutated genes in AML to establish the biological role of each mutation.

The molecular characterization of the 700 samples which are estimated to pick up during the project will consist of massive sequencing of genes recurrently mutated in AML (ASXL1, had, CBL, CEBPA, DNMT3A, EZH2, FLT3, GATA2, IDH1, IDH2, JAK2, KIT, KRAS, MPL, MLL, NPM1, NRAS, PTPN11, RUNX1, SETBP1, SF3B1, SRSF2, TET2, TP53, U2AF1, WT1). Found mutations will be collated in the different databases of somatic variations to establish which of them could be classified as a driver or passenger.

DETAILED DESCRIPTION:
All patients diagnosed with AML (new diagnosis or relapsed/refractory disease) can be included.

This project aims to establish a platform for comprehensive diagnostic and research platform in the context of the Spanish PETHEMA cooperative group, constituted by 80 institutions and seven central laboratories with extensive technological capacity.

This will be a prospective, multicenter, non-interventional study. It will be performed in 7 central laboratories (Hospital Universitario la Fe, Hospital Universitario de Salamanca, Hospital 12 de Octubre, Hospital Universitario Virgen del Rocío, Hospital Reina Sofía, Hospital Dr. Negrín and Clínica Universidad de Navarra) from the spanish PETHEMA group that will receive and process bone marrow and peripheral blood samples from AML patients at diagnosis and at resistance or first and subsequent relapses. In parallel, all patients will be enrolled in the ongoing PETHEMA epidemiologic registry of AML with a large number of clinical data however no safety information/Adverse Events about drug treatments will be collected. Currently, the PETHEMA group is reporting 600 newly diagnosed patients per year and accounts for 5000 cases in the data-base.

It is expected that the investigator will analyze 450 samples from 450 newly diagnosed patients that will participate in this study in a period of 2 years (225 per year). This means that roughly 40% of all AML patients from the PETHEMA group institutions will be included in the study.

In addition, other 250 samples from relapsing/refractory patients will be included in 2 years. Of these 250 samples form relapsing/refractory patients, it is expected that 150 samples will be drawn from patients in whom the sample was already analyzed at diagnosis in the current study, and 100 samples will be drawn form 100 additional patients that were not previously included in the study at the initial diagnosis. So, the expected distribution of analyzed samples will be: 450 at diagnosis, 150 resampling at first relapse from patients already analyzed at diagnosis, and 100 samples at first or subsequent relapse from patients not included in the study at the time of diagnosis. The investigator expect at least 500 patients and 700 samples.

Molecular diagnosis by NGS will be rapidly reported to the treating physician (<48-72 hours), in order to facilitate inclusion of patients in potential targeted therapy trials in AML.

Through the analysis of leukemic cells in samples from a large cohort of patients treated homogeneously, it is intended to delve into the prognostic value of genetic lesions that are observed at diagnosis by means of a large panel of mutations by next-generation sequencing. Thanks to this ambitious cooperative study, the investigator will be in an unprecedented and novel situation to understand the cellular mechanisms associated with chemoresistance of leukemic cells. This could allow us to design new therapeutic strategies of personalized medicine that will be able to eradicate these cells with minimal toxic effects on patients with AML.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients (≥18 years) with AML (excluding APL) according to the WHO criteria (2008), regardless of the treatment administered by their treating physician.
* Patient has to sign the informed consent form, allowing for sampling, analyses and reporting of the mutational results.
* AML at diagnosis and at relapse or refractoriness.

Exclusion Criteria:

* Genetic diagnosis of acute promyelocytic leukemia
* No Informed Consent Form

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients (≥18 years) with AML (excluding APL) according to the WHO criteria (2008), regardless of the treatment administered by their treating physician
Sampling Method: Non-Probability Sample
Enrollment: 900 (Actual)
Dates: Start 2017-10-06 (Actual); Primary Completion 2019-10-15 (Actual); Study Completion 2019-10-15 (Actual)

PRIMARY OUTCOMES:
Molecular diagnosis of acute myeloid leukemia | 3 years
  To develop a Spanish nationwide diagnostic platform to perform centralized and standardized rapid molecular diagnosis by next generation sequencing (NGS) in patients diagnosed with AML.
  NGS studies will be done in stem cell leukemic population. The analysis of the samples to the diagnosis will be carried out using the 26 consensus genes: ASXL1 had, CBL, CEBPA, DNMT3A, EZH2, FLT3, GATA2, IDH1, IDH2, JAK2, KIT, KRAS, MPL, MLL, NPM1, NRAS, PTPN11, RUNX1, SETBP1, SF3B1, SRSF2, TET2, TP53, U2AF1, WT1. Regarding the 26 genes panel, it would have the advantage that the quantification of DNA from each sample will be carried out by fluorimetry using the AmpliSeq or TruSeq on Ion platforms torrent Proton or MySeq are handled in different laboratories. Using NGS techniquesthe investigator will detect the recurrently mutated genes in AML to establish the biological role of each mutation.

CONTACTS AND LOCATIONS:
Overall Officials: Pau Montesinos, Dr, Principal Investigator — PETHEMA Foundation
Locations (7):
- Spain (7):
  - Hospital Reina Sofía, Córdoba
  - Hospital Dr. Negrín, Las Palmas de Gran Canaria
  - Hospital 12 de Octubre, Madrid
  - Clínica Universidad de Navarra, Pamplona
  - Hospital General Universitario, Salamanca
  - Hospital Virgen del Rocío, Seville
  - Hospital Universitari i Politècnic La Fe, Valencia

IPD SHARING:
Plan to Share IPD: No